CLINICAL TRIAL: NCT05340270
Title: PD-1 Inhibitor Plus GP Chemotherapy as Neoadjuvant Therapy for Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase II, Multicenter, Randomized Controlled Clinical Trial
Brief Title: PD-1 Inhibitor Plus GP as Neoadjuvant Therapy for Locoregionally Advanced Nasopharyngeal Carcinoma
Acronym: NeoTurbo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Collaborators: Hainan People's Hospital (Other); Wuzhou Red Cross Hospital (Other); First People's Hospital of Yulin (Other); Fourth Affiliated Hospital of Guangxi Medical University (Other); Guigang People's Hospital (Other); LiuZhou People's Hospital (Other); Afﬁliated Hospital of North Sichuan Medical College (Other)
Responsible Party: Principal Investigator, Kai Hu, professor, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangxiMUHK2
Record Dates: First submitted 2020-03-19; First posted 2022-04-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma; Neoadjuvant Therapy; PD-1 Inhibitor
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor + GP Group (Experimental): PD-1 inhibitor plus GP chemotherapy as Neoadjuvant Therapy followed by IMRT combined with cisplatin concurrent chemotherapy
  Interventions: Drug: PD-1 inhibitor+GP
- GP Group (Active Comparator): GP chemotherapy as Neoadjuvant Therapy chemotherapy followed by IMRT combined with cisplatin concurrent chemotherapy
  Interventions: Drug: GP

INTERVENTIONS:
Drug: PD-1 inhibitor+GP — PD-1 inhibitor (200-240mg), gemcitabine (1000mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1) every three weeks for three cycles as neoadjuvant therapy, then followed by IMRT and cisplatin (100mg/m2, d1, 22, 43 of RT) during concurrent chemoradiotherapy.
  Arms: PD-1 inhibitor + GP Group
Drug: GP — Gemcitabine (1000mg/m2 on day 1,8) and cisplatin (80mg/m2 on day 1) every three weeks for three cycles as neoadjuvant therapy, then followed by IMRT and cisplatin (100mg/m2, d1, 22, 43 of RT) during concurrent chemoradiotherapy.
  Arms: GP Group

SUMMARY:
The purpose of this Phase II, Multicenter, Randomized Controlled Clinical Trial is to evaluate the efficacy and safety of PD-1 inhibitor Plus GP chemotherapy as Neoadjuvant Therapy in the Treatment of Locoregionally Advanced Nasopharyngeal Carcinoma.

DETAILED DESCRIPTION:
Induction chemotherapy plus concurrent chemoradiotherapy has the IIA evidence and the gemcitabine plus cisplatin (GP) regimen has the I evidence in the National Comprehensive Cancer Network (NCCN) guidelines for the treatment of locoregionally advanced nasopharyngeal carcinoma (NPC). More and more evidence shows that immunotherapy combined with chemotherapy has a synergistic effect in treating tumors. GP chemotherapy combined with PD-1 inhibitor has achieved the initial effect in NPC. With the development of radiotherapeutic techniques and equipment as well as advances in treatment modalities, the 5-year overall survival of patients with non-disseminated NPC has exceeded 80%. But there are still about 20-30% of NPC patients who experienced recurrence or metastasis after radical chemoradiotherapy, especially locoregionally advanced patients. In order to improve their survival, we conduct this clinical trial to determine whether GP chemotherapy combined with PD-1 inhibitor as neoadjuvant therapy can improve the failure-free survival rate of locoregionally advanced NPC patients and provide new evidence for their neoadjuvant therapy of them.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma(WHO II/III).
2. Original clinical staged as T4NanyM0 or TanyN2-3M0 (according to AJCC 8th edition), with no evidence of distant metastasis.
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L, and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤1.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Age > 65 or < 18.
2. Receiving radiotherapy or chemotherapy or targeted therapy or immunotherapy previously.
3. Severe cerebrovascular disease/canker/psychosis.
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients who received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
6. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
7. Suffering from active infection diseases and in need of treatment.
8. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
9. Pregnant or breastfeeding.
10. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer and papillary thyroid carcinoma.
11. Has known allergy to large molecule protein products or any compound of PD-1 antibody.
12. Has a known history of the human immunodeficiency virus (HIV) infection.
13. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-03-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | up to 24 months
  the time from registration to treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Complete Response (CR) | up to 9 weeks
  the complete disappearance of the target and non-target lesion identified at baseline after radiological evaluation by MRI. Disease response was evaluated after the completion of the neoadjuvant therapy, according to RECIST 1.1.
Overall survival | up to 24 months
  the time from registration to death due to any cause, or censored at date last known alive.
Locoregional failure-free survival(LRRFS) | up to 24 months
  the time from registration to the first locoregional relapse or death from any cause.
Distant metastasis-free survival(DMFS) | up to 24 months
  the time from registration to the first distant metastasis or death from any cause.
Adverse events (AEs) | up to 24 months
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Quality of life（QOL） | up to 24 months
  Assessed by European Organization for Research and Treatment of Cancer's quality of life questionnaire(QLQ)-C30

CONTACTS AND LOCATIONS:
Overall Officials: RENSHENG WANG, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided